CLINICAL TRIAL: NCT07124923
Title: Effectiveness of a Continuous Care Intervention by the Endocrinology and Nutrition Service in Primary Care to Improve the Control of Type 2 Diabetes Mellitus in Terres de l'Ebre, Catalonia
Brief Title: Continuous Care Intervention in Primary Care to Improve Type 2 Diabetes Control in Terres de l'Ebre, Catalonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Collaborators: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); Institut Catala de Salut (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 009/2024; 2024 DI 00039 (Other: AGAUR. Agència de Gestió d'Ajuts Universitaris i de Recerca)
Record Dates: First submitted 2025-07-16; First posted 2025-08-15 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus Type 2
Keywords: HbA1c; Primary Care; Continuity of Care; Training
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will maintain blinding for participating patients, the data manager, the principal investigator, the statistician and the rest of the research team members. However, the primary care professionals who will receive the intervention, the trainers, those responsible for data extraction and the members of the training committee will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuity-of-Care Training for Primary Care Professionals (Experimental): A parallel-group randomized clinical trial will be conducted in 11 primary care centers of the Terres de l'Ebre area (Catalan Health Institute). Randomization was performed by the data extractor before pseudonymization using simple randomization (1:1 ratio), generating values 0 and 1. Centers scoring <0.5 were assigned to the control group; those ≥0.5 to the intervention group, resulting in 5 intervention and 6 control centers.
  Interventions: Other: Continuity-of-Care intervention
- Usual Care (No Continuity-of-Care Training) (No Intervention): Primary care professionals provide care according to current local standard practices without receiving specific training on continuity-of-care strategies.

INTERVENTIONS:
Other: Continuity-of-Care intervention — The intervention is a structured, multidisciplinary training and feedback program led by the Endocrinology Service at HTVC in collaboration with primary care centers in Terres de l'Ebre.
  Four endocrinologists and four nurses (three educators and one diabetic foot referent) will provide onsite training to primary care physicians and nurses. Training includes six modules with theoretical and practical components, covering T2DM management, cardiovascular risk reduction, and diabetic foot care. Sessions will be held biweekly and delivered by doctor-nurse teams rotating through the participating primary care centers from July 2025 to July 2026, with each center receiving a total of 15 sessions per year.
  The program also includes regular feedback to professionals on clinical performance and patient outcomes, adapting content to each center's needs. A qualitative component, involving focus groups before and after the intervention, will gather feedback and inform future implementation.
  Arms: Continuity-of-Care Training for Primary Care Professionals

SUMMARY:
This randomized, parallel-group clinical trial evaluates the effectiveness of a continuity of care intervention to improve metabolic control in adults with type 2 diabetes mellitus (T2DM) in the Terres de l'Ebre health region. The intervention, led by the Endocrinology Service at Hospital de Tortosa Verge de la Cinta (HTVC), involves structured, multidisciplinary training and feedback provided by endocrinologists and nurse educators to primary care professionals. Training modules combine theoretical and practical content focused on current diabetes management.

Primary care centers are randomized to intervention or control arms. Eligible participants are adult patients with an active diagnosis of T2DM for at least 12 months as of January 2025, registered in the eCAP system. All primary care professionals in intervention centers participate in the training.

The intervention is conducted over one year (July 2025-July 2026). Outcomes are assessed at baseline, 6, 12, and 24 months. The primary outcome is HbA1c; secondary outcomes include other health indicators, professional knowledge and engagement, and organizational variables. A qualitative component gathers professional input before and after the intervention to inform future implementation. All data are anonymized to ensure confidentiality.

DETAILED DESCRIPTION:
T2DM is a highly prevalent chronic disease, accounting for approximately 90% of all diabetes cases, and is primarily managed in the primary care setting. The complexity of optimizing metabolic control in T2DM has increased, as current guidelines recommend a multifactorial approach that addresses not only glycemic control but also cardiovascular risk and multimorbidity. Glycosylated hemoglobin (HbA1c) remains the principal marker for assessing glycemic control and predicting diabetes-related complications.

Despite the availability of evidence-based clinical practice guidelines, their implementation in routine care is often suboptimal due to factors such as limited time, resources, clinical inertia, and challenges with patient adherence. Interventions targeting healthcare professionals and organizational processes-such as structured training, audit and feedback, and system-level changes-have shown promise in improving metabolic outcomes, particularly among patients with suboptimal glycemic control.

This study is a randomized, parallel-group clinical trial designed to evaluate the effectiveness of a continuity of care intervention led by the Endocrinology Service at HTVC, in collaboration with primary care centers in the Terres de l'Ebre health region. Primary care centers will be randomized to either the intervention or control group.

The intervention consists of structured, multidisciplinary training and feedback provided by endocrinologists and nurse educators to primary care physicians and nurses. Training sessions are delivered in modules that combine theoretical and practical content, with a focus on up-to-date diabetes management strategies and the needs of each primary care center. The endocrinology team includes endocrinologists, nurse educators, and a specialist nurse from the Diabetic Foot Unit. Training will be delivered onsite at intervention centers in scheduled sessions over a one-year period.

A qualitative component is integrated into the study, involving focus groups with participating primary care professionals before and after the intervention. This aims to gather insights on professional perspectives, identify barriers and facilitators, and inform the adaptation and future implementation of the intervention.

The primary outcome is improvement in HbA1c, with secondary outcomes including additional patient health indicators, professional knowledge and engagement, and organizational variables. Data collection will occur at baseline, 6, 12, and 24 months. All data will be anonymized to ensure confidentiality.

This study aims to provide evidence on the effectiveness of a multidisciplinary, continuity of care intervention in improving metabolic control for adults with T2DM in a real-world primary care setting.

ELIGIBILITY:
Inclusion Criteria:

Enrollment will begin in July 2025, aligned with the initiation of training sessions for healthcare professionals (physicians and nurses).

Eligible participants must:

* Be adults (≥18 years old)
* Have an active diagnosis of T2DM documented in the eCAP primary care electronic health record system
* Have a duration of T2DM of at least 12 months as of January 2025

Exclusion Criteria:

* Diagnosis of type 1 diabetes mellitus (T1DM)
* T2DM managed by a specialist at the time of inclusion
* Current treatment with systemic corticosteroids
* Active neoplasia (malignancy)
* Gestational diabetes
* Pregnancy or breastfeeding
* Diagnosis of MACA (advanced chronic disease with life expectancy <1 year)
* Complex chronic patients (CCP)
* Diagnosis of dementia
* Institutionalized patients or those residing in social healthcare facilities
* Age over 90 years
* Age under 18 years
* Severe psychiatric illness (e.g., psychosis, bipolar disorder, major depression)
* History of kidney transplant
* Undergoing dialysis
* History of alcohol or drug abuse

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7792 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
HbA1c | At enrollment, 6, 12, and 24 months after enrollment.
  Evaluate the percentage improvement in HbA1c levels in relation to healthcare professionals' attendance at training sessions.

SECONDARY OUTCOMES:
Change in total cholesterol and LDL cholesterol | At enrollment, 6, 12, and 24 months after enrollment.
  Mean change in total and LDL cholesterol levels from baseline, measured in mg/dL.
Change in systolic and diastolic blood pressure | At enrollment, 6, 12, and 24 months after enrollment.
  Mean change in systolic and diastolic blood pressure from baseline, measured in mmHg.
Change in smoking status | At enrollment, 6, 12, and 24 months after enrollment.
  Change in smoking status (current, former, never) and number of cigarettes smoked per day.
Change in Body Mass Index (BMI) | At enrollment, 6, 12, and 24 months after enrollment.
  Mean change in BMI (Kg/m2) from baseline. BMI will be calculated as weight in kilograms divided by height in meters squared.
Percentage of participants adherent to screening protocol for T2DM complications | At enrollment, 6, 12, and 24 months after enrollment.
  Percentage of participants who complete all recommended screenings for chronic complications of T2DM, including screening for retinopathy, nephropathy, foot examination, and cardiovascular assessment.
Referrals to the Diabetic Foot Unit | At enrollment, 6, 12, and 24 months after enrollment.
  Evaluate the association between attendance at diabetic foot training and referrals to the Diabetic Foot Unit.
Emergency assistance for metabolic decompensations | At enrollment, 6, 12, and 24 months after enrollment.
  Evaluate whether patients present to emergency care with a diagnosis of metabolism and nutrition disorder according to CIE-10 ( CIE-10 E00-E90)
Number of hospital referrals from primary care | At enrollment, 6, 12, and 24 months after enrollment.
  Evaluate the number of hospital referrals to endocrinology specialty consultation after primary care attendance.
Medication changes | At enrollment, 6, 12, and 24 months after enrollment.
  Assess the association between professional attendance at training and medication changes.
Number of patient visits to primary care | At enrollment, 6, 12, and 24 months after enrollment.
  Evaluate the number of patient visits to primary care, stratified by nursing and physician attendance.
Professional perceptions of relevance, feasibility and impact of the Continuity-of-Care intervention | Pre-intervention and 1 month post-intervention
  Professional perceptions of the Continuity-of-Care intervention will be assessed through pre- and post-intervention focus groups. Focus groups will be conducted with professionals from different disciplines (primary care doctors and nurses). Transcripts will be analyzed using thematic content analysis to assess perceptions of relevance, feasibility, and impact of the intervention.
Professional experiences with implementing the Continuity-of-Care intervention, including perceived barriers and facilitators | Pre-intervention and 1 month post-intervention.
  Professional experiences with implementing the Continuity-of-Care intervention will be assessed through pre- and post-intervention focus groups. Focus groups will be conducted with professionals from different disciplines (primary care doctors and nurses). Transcripts will be analyzed using thematic content analysis to assess experiences related to implementation and perceived barriers/facilitators.

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Miret Llauradó, MD, Principal Investigator — Catalan Institute of Health
Locations (12):
- Spain (12):
  - Abs Amposta, Amposta, Tarragona
  - Abs Deltebre, Deltebre, Tarragona
  - Abs Ametlla-Perelló, El Perelló, Tarragona
  - ABS FLIX, Flix, Tarragona
  - Abs Gandesa, Gandesa, Tarragona
  - Abs Ampolla-Aldea, L'Ampolla, Tarragona
  - Abs Mora La Nova, Móra la Nova, Tarragona
  - Abs La Ràpita-Alcanar, Sant Carles de la Ràpita, Tarragona
  - Abs Tortosa Est, Tortosa, Tarragona
  - Abs Tortosa Oest, Tortosa, Tarragona
  - Hospital de Tortosa Verge de la Cinta, Tortosa, Tarragona
  - Abs Ulldecona, Ulldecona, Tarragona

IPD SHARING:
Plan to Share IPD: No
Data sharing will be upon request directly to the Principal Investigator.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-07-20): https://cdn.clinicaltrials.gov/large-docs/23/NCT07124923/Prot_SAP_ICF_000.pdf